CLINICAL TRIAL: NCT04933929
Title: Personalized Dietary Advice 3 Months After Discharge From Hospitalization in Geriatrics: Effect on Nutritional Status According to Coronavirus Disease 2019 (Covid-19) Status (Positive or Negative) During Hospitalization
Acronym: COVINUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gérond'if (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-A02168-31
Record Dates: First submitted 2021-05-24; First posted 2021-06-22 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2)
Keywords: Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2)-positive patients; Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2)-negative patients; Coronavirus disease 2019 (COVID-19)
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Post-hospitalization nutritional monitoring, carried out by dieticians from Saveurs & Vie. Consultations are done remotely, by phone only. Dietitians have gained experience in home nutritional monitoring of elderly people over the phone during the first wave of Coronavirus disease 2019 (COVID-19) .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coronavirus disease Positive group "Covid (+)" (Experimental): Positive PCR test.
  Interventions: Behavioral: Post-hospitalization nutritional monitoring
- Coronavirus disease Negative group "Covid (-)" (Active Comparator): Negative PCR test.
  Interventions: Behavioral: Post-hospitalization nutritional monitoring

INTERVENTIONS:
Behavioral: Post-hospitalization nutritional monitoring — Post-hospitalization nutritional monitoring, carried out by dieticians from Saveurs & Vie. Consultations are done remotely, by phone only. Dietitians have gained experience in home nutritional monitoring of elderly people over the phone during the first wave of Coronavirus disease 2019 (COVID-19) .

SUMMARY:
The principal aim of this interventional, multicentre study is to compare the impact of a follow-up by monthly telephone dietetic consultations, started 3 months after discharge from hospital, for a period of 3 months, on the energy intake in patients elderly people recently hospitalized for Coronavirus disease 2019 (Covid-19), Coronavirus disease Positive group "Covid (+)", or not, Coronavirus disease Negative group"Covid (-)".

The main outcome measure is to compare the total energy intake at 6 months, after 3 months of dietary consultations, between Coronavirus disease Positive group "Covid (+)" and Coronavirus disease negative group "Covid (-)".

DETAILED DESCRIPTION:
This study consists of nutritional monitoring after hospitalization, carried out by dieticians. Consultations are done remotely, by phone only.

Eligible subjects are included, either upon discharge from hospital or within 3 months (at the latest) following their hospitalization.

135 subjects will be included, 50% will be included in Coronavirus disease Positive group "Covid (+)" and 50% in the Coronavirus desease negative group "Covid (-)" .

The following data will be collected

* At Inclusion (D0): Average length of hospital stay, medical diagnoses, severity of hospital stay, autonomy and dependency scores, albumin and body mass index (BMI).
* At M3, M4, M5 and M6: Dietary monitoring data, patient's vital status and dependency scores.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized or having been hospitalized in acute geriatrics
* Living at home 3 months after hospitalization in acute geriatrics
* Having a good understanding of the French language
* Being able to understand the study information and participate in telephone follow-up
* Having read the information notice and agreeing to participate in the study
* For the Covid (+) group: hospitalized for Covid-19 (diagnostic confirmation by positive RT-PCR)
* For the Covid group (-): hospitalized for any other reason (negative RT-PCR)

Exclusion Criteria:

* Patient refusing to participate in the study
* Subject to a legal protection measure (curatorship, guardianship or safeguard of justice)
* With cognitive impairment making it impossible to understand the study protocol and express consent.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2021-04-22 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Comparison of total energy requirements, after 3 months of dietary consultations, between Covid (+) and Covid (-) groups. | 6 months
  A 30 to 40 minute telephone survey by a dietitian, with:
  * the reminder of food intake over 24 hours, estimation of the weight of each food and quantification in kcal / day and grams of protein / day.
  * This assessment of food intake will be followed by nutritional advice adapted to the severity of undernutrition, spontaneous food intake, the subject's tastes and dislikes, and the possibilities of preparing the necessary dishes and textures.

SECONDARY OUTCOMES:
Assessment of the degree of patient dependence according "Index of Independence in Activities of Daily Living" KATZ scale | At inclusion
  This is a measurement of the subject's ability to perform activities of daily living independently without including minimum and maximum values
Assessment of patient's level of dependence through an appreciation of instrumental activities of daily living according Lawton scale | At inclusion
  Assessment of older people: Self-maintaining and instrumental activities of daily living without including minimum and maximum values
Comparison of weight variation by measuring the Body Mass Index (BMI) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Agathe RAYNAUD-SIMON, MD PhD, Study Chair — Geriatric Department, Bichat, Beaujon and Bretonneau hospitals
Locations (1):
- Geriatric Department, Bichat, Beaujon and Bretonneau hospitals, Paris, IIe-de-France, France